CLINICAL TRIAL: NCT04243694
Title: Sustainable Mindfulness and Resilience Training (SMART)
Acronym: SMART
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Reduction in funding.
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 19-27771
Record Dates: First submitted 2019-10-07; First posted 2020-01-28 (Actual); Last update posted 2021-01-20 (Actual); Status verified 2021-01

CONDITIONS: Caregiver Stress; Autism Spectrum Disorder
Keywords: caregiver stress; caregiver; parent; asd; autism; autism spectrum disorder
MeSH Terms: conditions — Caregiver Burden; Autism Spectrum Disorder; Child Development Disorders, Pervasive; Autistic Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): mindfulness intervention administered
  Interventions: Behavioral: Mindfulness training
- Control group (No Intervention): no intervention administered

INTERVENTIONS:
Behavioral: Mindfulness training — Participants of the intervention group will receive 6-weeks of mindfulness training.
  Arms: Intervention group

SUMMARY:
Investigators are proposing a 6-week mindfulness and resilience training intervention tailored for caregivers of children with autism. Investigators will assess increases the caregiver's well-being and levels of psychological acceptance of their life situation as it relates to their child with autism. The mindfulness training focuses on self-regulation of emotional responses and acceptance of internal experiences. Self-report measures and qualitative interviews will be administered at baseline and post-intervention. Investigators will compare the active group to a control group of caregivers who are on the waitlist to receive the intervention.

DETAILED DESCRIPTION:
Investigators will prospectively examine a sample comprised of parental caregivers (ages 20 to 60) of children with autism spectrum disorder (ages 3 to 12) to determine how responses to the chronic stress of caregiving may contribute to psychological distress (e.g depression, caregiving burden, self-reported sleep).

All participants:

Participants will be randomized into the active group vs. wait list control group. Investigators will assess indices of psychological health at 2 time points over 6 weeks (length of intervention) - a Baseline Assessment, and a Follow-up Assessment. Both baseline and follow-up assessments include the same battery of questionnaires.

Daily/nightly diaries will also be completed by participants in the 7 days leading up to the baseline and follow-up time points.

In addition to self-report measures, investigators will conduct a 20-25 minute qualitative interview with caregivers both pre and post-intervention. The interview is optional and will be conducted via telephone before beginning the six-week course and within two weeks of finishing the course. The interview will be used to assess caregiver's acceptance of their child's condition and better understand their personal perception of their own acceptance. Interviews questions will be open-ended and may be modified based on the caregiver's response. An example question includes, "How hard has it been to accept your child has ASD?

Control group only:

The control group will be waitlisted and enrolled in the next 6-week mindfulness course. Investigators expect the next mindfulness course for the waitlist control group to be held within 1-3 months of the initial active group course.

Active group only:

The active group will participate in a mindfulness resilience training intervention. The intervention consists of weekly 2 hour classes held at UCSF Parnassus Campus over the course of 6 weeks. The study PI, Dr. Elissa Epel, will lead the intervention classes teaching the fundamentals of mindfulness training. The training focuses on acceptance and awareness of the present moment.

ELIGIBILITY:
Inclusion Criteria:

* Age 20-60 years old
* Full time caregiver for a child with ASD, aged 3 to 12
* Child diagnosed with ASD for a minimum of 6 months
* English Speaking

Exclusion Criteria:

* Any conditions that may make it difficult to participate in a mindfulness group (e.g., psychotic disorder, personality disorder)

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2020-07-01 (Actual); Study Completion 2020-07-01 (Actual)

PRIMARY OUTCOMES:
Acceptance of child's diagnosis: Acceptance of Diagnosis of Autism-modified scale | 6 weeks
  Measured by the Acceptance of Diagnosis of Autism-modified scale (example item "I have a greater acceptance of my child's challenges than I used to.")
Acceptance of one's negative experiences (experiential avoidance, negative emotions and thoughts): Acceptance and Action Questionnaire | 6 weeks
  Measured by the Acceptance and Action Questionnaire (example item rating on a scale "I'm afraid of my feelings", the Brief Experiential Avoidance Questionnaire (measures intentional avoidance of thoughts, feelings and experiences associated with distress), and the Self Compassion Scale (measures the degree to which individuals display self-kindness against self-judgment, common humanity versus isolation, and mindfulness versus over-identification).
Acceptance of one's momentary situation as assessed by daily mind states (mind wandering, rejection vs. engagement in current moment): daily diary assessments | 6 weeks
  Measured by daily diary assessments

CONTACTS AND LOCATIONS:
Overall Officials: Elissa Epel, PhD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No